CLINICAL TRIAL: NCT07078682
Title: An Open-Label, Single-Group Study to Evaluate the Effect of Elix Cycle Balance & Elix Daily Harmony on Fibroid-related Symptoms
Brief Title: An Open-Label Study to Evaluate the Effect of Elix Cycle Balance & Elix Daily Harmony on Fibroid-related Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zenchi, Inc. (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20790
Record Dates: First submitted 2025-07-11; First posted 2025-07-22 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Uterine Fibroids; Leiomyoma; Menstrual Pain
MeSH Terms: conditions — Leiomyoma; Dysmenorrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elix Cycle Balance & Elix Daily Harmony (Experimental): Participants will receive two investigational herbal supplements daily for 24 weeks.
  Interventions: Dietary Supplement: Elix Daily Harmony

INTERVENTIONS:
Dietary Supplement: Elix Daily Harmony — Each morning, 1-2 hours after their first meal, they will mix the following into room-temperature or warm water and consume:
  Elix Daily Harmony: 3 droppers full (approximately 2.5 mL) Elix Cycle Balance: 6 droppers full (approximately 5.0 mL)

SUMMARY:
This is a 24-week, single-arm, open-label, virtual study evaluating the effects of Elix Cycle Balance and Elix Daily Harmony on uterine fibroid-related symptoms and quality of life in 42 participants. Participants will self-administer the investigational herbal supplements daily and complete validated questionnaires at scheduled timepoints to assess symptom severity and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Be female.
* Be aged 20-45.
* BMI 18.5 - 24.9 kg/m2
* Self-reported prior diagnosis of uterine fibroids.
* Anyone who is generally healthy - does not live with any uncontrolled chronic disease.
* Self-reported moderate to severe discomfort during menstruation, related to pelvic cramps, bloating, mood swings, or fatigue.
* Self-reported menstrual cramps during their cycle, for the past six months minimum.
* If taking hormonal birth control, has been doing so consistently for at least three months, and experiences a menstrual cycle with a period.
* If taking other oral over-the-counter supplements or herbal remedies, has been consistently taking these for at least three months prior to starting the study, and is willing to maintain this routine for the study duration.
* Willing to refrain from introducing any products or any new forms of medication or supplements for the study duration.
* Willing to refrain from any other dietary supplements or herbal remedies targeting the menstrual cycle during the study period.
* Willing to refrain from any new vaccines during the 6 month period.
* Follows a stable, consistent exercise regimen and are willing, for the duration of the study, to not decrease or increase the amount of exercise in their regimen.
* Agrees to refrain from any lifestyle changes that may affect their menstrual cycle for the duration of the study (for example, getting on or off hormonal birth control, reducing the amount of exercise).
* If using any other interventions, such as massage, chiropractic medicine, or acupuncture, agrees not to increase or decrease the number of these other interventions during the study period.
* Resides in the United States.

Exclusion Criteria:

* Does not experience a regular menstrual cycle (21-35 days).
* Does not experience menstrual cramping.
* Follows an extreme diet intervention such as dry fasts, water fasts, or ketogenic diets.
* Anyone who has experienced significant weight loss in the past three months prior to study participation.
* Unwilling to stop the use of any medication or herbal remedies/supplements that can affect the menstrual cycle.
* Anyone with pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Anyone with known severe allergic reactions.
* Anyone with any allergies or sensitivities to any of the study product ingredients.
* Any women who are pregnant, breastfeeding, or trying to conceive (or who will be at any point during the study period).
* Anyone unwilling to follow the study protocol.
* Has stopped, started, or changed hormonal birth control in the past three months.
* Previous users of Elix Cycle Balance.
* Anyone who is currently a smoker or has been a smoker in the past 3 months.
* Anyone who has been diagnosed with the following conditions: PCOS, Endometriosis, PMDD, Adenomyosis, Hashimoto's thyroiditis, Grave's disease (and any other thyroid disorders), hyperprolactinemia, Cushing's disease, congenital adrenal hyperplasia, anorexia, bulimia, orthorexia, binge eating, any other eating disorder.
* History of endocrine disorders such as thyroid disorder, Type 1 or 2 diabetes, or other.
* History of hypertension, hyperlipidemia, or previous venous embolism.
* Overweight/obesity (BMI > 25 kg/m2).
* Women with other causes of chronic pelvic pain, including infectious disease, gastrointestinal, psychological disorders, fibromyalgia, and chronic fatigue syndrome.
* Hysterectomy, myomectomy, or bilateral salpingo-oophorectomy or other gynecological medical or surgical treatment in the last 6 months.
* History of an abnormal pap smear.
* History of neoplasia of gynecological origin and/or existence of uterine malformations.
* Chronic urinary tract infections or diagnosed functional gastrointestinal conditions like IBS, IBD, Crohn's disease, or ulcerative colitis.
* Currently partaking in another research study or will be partaking in any other research study for the next 24 weeks, or at any point during this study's duration.
* Consume more than 5 alcoholic drinks per week
* Had a vaccine in the last 3 months

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in uterine fibroid-related symptom severity | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
  Measured as change in menstrual pain and bleeding volume using the validated Uterine Fibroid Symptom Health-Related Quality of Life Questionnaire (UFS-QOL) total and subscale scores.

SECONDARY OUTCOMES:
Change in fibroid-related health-related quality of life domains | Baseline, Week 4, Week 8, Week 12, Week 16, Week 20, and Week 24
  Measured as change in self-reported scores on UFS-QOL and study-specific questions addressing energy levels, emotional well-being, self-consciousness, sleep quality, and limitations in daily and social activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No